CLINICAL TRIAL: NCT00798811
Title: Multicenter Clinical Trial to Evaluate Efficacy of High-dose Chemotherapy With Autologous Stem Cell Rescue for Children With High-risk Brain Tumors
Brief Title: High-dose Chemotherapy With Autologous Stem Cell Rescue in Pediatric High-risk Brain Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: KSPNO stem cell transpantation committee (Unknown)
Responsible Party: Ki Woong Sung, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-12-009
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Brain Tumor
Keywords: brain tumor; high-dose chemotherapy; autologous stem cell transplantation; infant
MeSH Terms: conditions — Brain Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- KSPNO-S-081 (Other): Reduced-dose Craniospinal Radiotherapy Followed by High-dose Chemotherapy and Autologous Stem Cell Rescue in Children with Newly Diagnosed High-risk Brain Tumor
  Interventions: Procedure: high-dose chemotherapy and autologous stem cell rescue
- KSPNO-S-082 (Other): High-dose Chemotherapy and Autologous Stem Cell Rescue in Infants and Young Children with Newly Diagnosed High-risk Brain Tumor To Avoid or Reduce Craniospinal Radiation
  Interventions: Procedure: high-dose chemotherapy and autologous stem cell rescue
- KSPNO-S-083 (Other): High-dose Chemotherapy and Autologous Stem Cell Rescue in Children with Recurrent Brain Tumor or Non-germinomatous Germ Cell Tumor with Inadequate Response to Conventional Treatment
  Interventions: Procedure: high-dose chemotherapy and autologous stem cell rescue

INTERVENTIONS:
Procedure: high-dose chemotherapy and autologous stem cell rescue — Surgery -> enroll Pre-RT chemotherapy (2 cycles: A1, B1) PBSC collection during first cycle (A1) (2nd look surgery if necessary) RT (Reduced dose CSI) Post-RT chemotherapy (4 cycles: A2, B2, A3, B3) (if relapse or progression prior to HDCT, off study -> enroll S-083 protocol) HDCT1 (CTE) HDCT2 (CM)
  Arms: KSPNO-S-081
Procedure: high-dose chemotherapy and autologous stem cell rescue — Surgery pre-HDCT chemotherapy (6 cycles: A1, B1, A2, B2, A3, B3) PBSC collection during first cycle of chemotherapy (A1) (2nd look surgery if necessary) (if relapse or progression prior to HDCT, off study -> enroll S-083 protocol) HDCT1 (CTE) HDCT2 (CM) (RT if necessary) Observe
  Arms: KSPNO-S-082
Procedure: high-dose chemotherapy and autologous stem cell rescue — (Surgery if possible) Chemotherapy (4 cycles) PBSC collection during first cycle of chemotherapy during 4th cycle of chemotherapy (if BM involvement) (RT, if possible, after PBSC collection) (if less than PR prior to HDCT, off study) HDCT1 (CTE) HDCT2 (CM)
  Arms: KSPNO-S-083

SUMMARY:
* Study No.: KSPNO-S-081 Reduced-dose Craniospinal Radiotherapy Followed by High-dose Chemotherapy and Autologous Stem Cell Rescue in Children with Newly Diagnosed High-risk Brain Tumor
* Study No.: KSPNO-S-082 High-dose Chemotherapy and Autologous Stem Cell Rescue in Infants and Young Children with Newly Diagnosed High-risk Brain Tumor To Avoid or Reduce Craniospinal Radiation
* Study No.: KSPNO-S-083 High-dose Chemotherapy and Autologous Stem Cell Rescue in Children with Recurrent Brain Tumor or Non-germinomatous Germ Cell Tumor with Inadequate Response to Conventional Treatment

DETAILED DESCRIPTION:
Although significant progress has been made in the treatment of brain tumors, the prognosis remains dismal in patients with relapsed tumor. The outlook for infants and young children is also poor, primarily because of the limited use of radiotherapy, although a recent report suggested that vigorous combination chemotherapy alone improved the survival of young children without macroscopic metastases at diagnosis. The prognosis is also not satisfactory when a large residual tumor remains after surgery or when leptomeningeal seeding is present at diagnosis. Given the above situation, we plan to explore the possible efficacy of high-dose chemotherapy and autologous stem cell rescue in patients with high-risk embryonal tumors, relapsed brain tumors and in infants and young children with brain tumors.High-dose chemotherapy and autologous stem cell rescue has improved the survival of children with high-risk solid tumors. this treatment strategy is based on the hypothesis that a dose escalation might improve the survival of children with high-risk solid tumors.Many investigators demonstrated that further dose escalation using sequential high-dose chemotherapy and autologous stem cell rescue might result in additional improvements in the survival of patients with high-risk tumors. As embryonal brain tumors are a chemosensitive tumors, a strategy using high-dose chemotherapy might be effective in the treatment of high-risk embryonal brain tumors and relapsed brain tumors. In addition, it might defer or eliminate irradiation in infants and young children with brain tumors

ELIGIBILITY:
Inclusion Criteria:

* KSPNO-S-081: newly diagnosed embryonal brain tumor, age >= 3 years
* KSPNO-S-082: all high-grade or malignant brain tumor, age <3 years
* KSPNO-S-083: recurrent embryonal brain tumors, recurrent CNS germ cell tumor

Exclusion Criteria:

* Patients with severe comorbid organ dysfunction (NCI grade > 2 organ toxicity) prior to high-dose chemotherapy
* Patients with progressed tumor prior to high-dose chemotherapy
* Patients whose parents do not want to undergo high-dose chemotherapy and autologous stem cell rescue

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
overall survival, event-free survival | one year

SECONDARY OUTCOMES:
toxicity | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Sung, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea